CLINICAL TRIAL: NCT04748458
Title: Retrospective Study About the Long-term Outcomes of Conical Tapered Stems in Cementless Total Hip Arthroplasty for Osteoarthritis Due to Congenital Hip Pathologies
Brief Title: Long-term Outcomes of Conical Tapered Stems in Cementless Total Hip Arthroplasty Due to Congenital Hip Pathologies
Acronym: RetroCone
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 589/2020/Oss/IOR
Record Dates: First submitted 2020-10-27; First posted 2021-02-10 (Actual); Results first posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2020-10

CONDITIONS: Dysplasia; Hip; Prosthesis Survival
MeSH Terms: conditions — Hip Dislocation; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Congenital hip pathologies: Conical tapered stem for osteoarthritis due to congenital hip pathologies
  Interventions: Device: Conical tapered stem

INTERVENTIONS:
Device: Conical tapered stem — Implantation of conical tapered stem

SUMMARY:
A retrospective consecutive population of patients treated with conical tapered stems in cementless total hip arthroplasty for osteoarthritis due to congenital hip pathologies will be selected. The aim of this retrospective study is to evaluate the long-term clinical and radiographic results of this implant and the survival rates in such a specific cohort.

DETAILED DESCRIPTION:
Congenital hip pathologies may severely alter the local anatomy of the hip, making total hip arthroplasty (THA) due to osteoarthritis after congenital hip pathologies challenging. While it seems that congenital hip pathologies did not significantly influence the outcomes when compared to THA after osteoarthritis, the choice of implant was demonstrated to impact the survival rates of the THA after congenital hip pathologies.

To date, no guidelines exist about the correct choice of hip implant in congenital hip pathologies: only mid-term case series are available. Conical tapered stems have been frequently suggested for the most difficult cases.

The aim of this study is to describe the survival rates and the long-term clinical and radiological outcome of conical tapered stems in THAs after congenital hip pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic hip osteoarthritis due to congenital hip pathologies
* Consecutive population with a minimum follow-up of 2 years
* Cementless total hip arthroplasty with conical tapered stem
* Pre-operative planning using CT
* Complete clinical and radiographic assessment

Exclusion Criteria:

* Other type of hip osteoarthritis
* Other type of implants
* Inadequate pre-operative planning (eg: no CT)
* Incomplete clinical and radiographic assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective, consecutive adult population treated with conical tapered stems in cementless total hip arthroplasty for osteoarthritis due to congenital hip pathologies.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Traina, Prof, Study Director — IRCCS Istituto Ortopedico Rizzoli, Bologna, ITaly
Locations (1):
- Chirurgia Protesica e dei Reimpianti di Anca e Ginocchio, IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Greber EM, Pelt CE, Gililland JM, Anderson MB, Erickson JA, Peters CL. Challenges in Total Hip Arthroplasty in the Setting of Developmental Dysplasia of the Hip. J Arthroplasty. 2017 Sep;32(9S):S38-S44. doi: 10.1016/j.arth.2017.02.024. Epub 2017 Feb 22. PMID 28291651
- [Result] Perry KI, Berry DJ. Femoral considerations for total hip replacement in hip dysplasia. Orthop Clin North Am. 2012 Jul;43(3):377-86. doi: 10.1016/j.ocl.2012.05.010. PMID 22819165
- [Result] Argenson JN, Flecher X, Parratte S, Aubaniac JM. Anatomy of the dysplastic hip and consequences for total hip arthroplasty. Clin Orthop Relat Res. 2007 Dec;465:40-5. doi: 10.1097/BLO.0b013e3181576052. PMID 17906591
- [Result] Pak P, de Steiger R. Cone femoral prosthesis for osteoarthritis of the hip with femoral dysplasia. J Orthop Surg (Hong Kong). 2008 Aug;16(2):206-10. doi: 10.1177/230949900801600216. PMID 18725674
- [Result] Taniguchi N, Jinno T, Koga D, Hagino T, Okawa A, Haro H. Cementless Hip Stem Anteversion in the Dysplastic Hip: A Comparison of Tapered Wedge vs Metaphyseal Filling. J Arthroplasty. 2017 May;32(5):1547-1552. doi: 10.1016/j.arth.2016.12.020. Epub 2016 Dec 22. PMID 28110848

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: hip
Period: Overall Study
Arm/Group | Congenital Hip Pathologies
Started | 85; 100 hip
Completed | 85; 100 hip
Not Completed | 0; 0 hip

BASELINE CHARACTERISTICS:
Units Other Than Participants: hip
Arm/Group | Congenital Hip Pathologies
Number analyzed (Participants) | 85
Number analyzed (hip) | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 85
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Italy | 85
Crowe I [Count of Units; unit: hip] — Hips classified according to the Crowe dislocation degree (scale from 1, minimal subluxation, to 4, high riding hip)
  hip | 46
Crowe II [Count of Units; unit: hip] — Hips classified according to the Crowe dislocation degree (scale from 1, minimal subluxation, to 4, high riding hip)
  hip | 30
Crowe III [Count of Units; unit: hip] — Hips classified according to the Crowe dislocation degree (scale from 1, minimal subluxation, to 4, high riding hip)
  hip | 14
Crowe IV [Count of Units; unit: hip] — Hips classified according to the Crowe dislocation degree (scale from 1, minimal subluxation, to 4, high riding hip)
  hip | 10

OUTCOME MEASURES:

1. Primary Outcome: Harris Hip Score
Description: Mean clinical results at last follow-up evaluated using the Harris hip score. Minimum-maximum values: 0-100. Best result: 100.
Time Frame: 15 months
Population: Total hip arthroplasties with a Wagner Cone implant in dysplasia
Measure: Mean (Standard Deviation); unit: points
Units Other Than Participants: hip
Arm/Group | Congenital Hip Pathologies
Number analyzed (Participants) | 85
Number analyzed (hip) | 100
points | 89.8 (6.8)

2. Primary Outcome: Survival Rate
Description: Percentage of survived implants (no component exchange or removed) described using Kaplan-Meier curve with 95% confidence interval. Minimum-maximum values: 0-100. Best result: 100.
Time Frame: 15 months
Population: Total hip arthroplasties with a Wagner Cone implant in dysplasia
Measure: Mean (95% Confidence Interval); unit: percentage of surviving hips
Units Other Than Participants: hip
Arm/Group | Congenital Hip Pathologies
Number analyzed (Participants) | 85
Number analyzed (hip) | 100
percentage of surviving hips | 98.9 [92.5 to 99.8]

3. Primary Outcome: Radiographic Cup Osseointegration
Description: Osseointegrated cups described using the Moore's criteria: the cup is osseointegrated when at least 3 criteria are present (radial trabeculae, superolateral buttress, inferolateral buttress, medial stress shielding, absence of radiolucent lines).
Time Frame: 15 months
Population: Total hip arthroplasties with a Wagner Cone implant in dysplasia
Measure: Count of Units; unit: hip
Units Other Than Participants: hip
Arm/Group | Congenital Hip Pathologies
Number analyzed (Participants) | 85
Number analyzed (hip) | 100
hip | 98

4. Primary Outcome: Radiographic Stem Osseointegration
Description: Osseointegrated stems described according to Engh's criteria
Time Frame: 15 months
Population: Total hip arthroplasties with a Wagner Cone implant in dysplasia
Measure: Count of Units; unit: hip
Units Other Than Participants: hip
Arm/Group | Congenital Hip Pathologies
Number analyzed (Participants) | 85
Number analyzed (hip) | 100
hip | 99

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Congenital Hip Pathologies
All-Cause Mortality (participants affected / at risk) | 4/85
Serious Adverse Events (participants affected / at risk) | 0/85
Other Adverse Events (participants affected / at risk) | 0/85

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT04748458/Prot_SAP_000.pdf